CLINICAL TRIAL: NCT07128069
Title: Can Vitamin D Reduce the Burden of COVID-19?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB20-0847
Record Dates: First submitted 2025-08-15; First posted 2025-08-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: vitamin D
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: 2,000-person two-arm, double-blinded randomized controlled trial, with half the subjects randomized to low dose vitamin D (400 IU/day), which will serve as the control group, and half to moderate dose vitamin D (4,000 IU/day)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose Vitamin D (400 IU/day) (Active Comparator): Subjects in this arm will be randomized to receive low dose vitamin D (oral, 400 IU/day) for 12 continuous months
  Interventions: Dietary Supplement: Vitamin D 400IU
- Moderate Dose Vitamin D (4000 IU/day) (Active Comparator): Subjects in this arm will be randomized to receive moderate dose vitamin D (oral, 4000 IU/day) for 12 continuous months
  Interventions: Dietary Supplement: Vitamin D 4000IU

INTERVENTIONS:
Dietary Supplement: Vitamin D 400IU — Low dose vitamin D (400 IU/day)
  Other Names: Vitamin D3
  Arms: Low Dose Vitamin D (400 IU/day)
Dietary Supplement: Vitamin D 4000IU — Moderate dose vitamin D (4000 IU/day)
  Other Names: Vitamin D3
  Arms: Moderate Dose Vitamin D (4000 IU/day)

SUMMARY:
The purpose of this study is to compare the risks of COVID-19 in individuals from the Chicagoland area and other communities in the United States randomized to low (400 IU/day) versus moderate (4,000 IU/day) dose vitamin D.

DETAILED DESCRIPTION:
This study will recruit 2,000 subjects from the Chicagoland area and across the United States to participate in the study from home. Subjects will be invited to volunteer to participate in the study through a variety of forms of outreach, mainly online (e.g., press releases, news interviews, social media, emails, etc.). The sample size was chosen to have at least 80% power to detect a 20% or larger decrease in the hazard of developing COVID-19 between study arms at p<0.05, based on an estimated monthly incidence of COVID-19 (3%/month for Black/Latinx persons and 1%/month for White persons) and an estimated fraction of persons already immune but unaware they have had COVID-19 (≤10%).

Subjects will take a daily dose of vitamin D and answer surveys about COVID-19 diagnosis and symptoms over 12 months after enrollment.

Our overall aim is to compare the risks of COVID-19 in adults at increased risk of COVID-19 randomized to low (400 IU/day) versus moderate (4,000 IU/day) dose vitamin D. Our specific aims are:

Aim 1: To compare the risk of developing COVID-19 in adults at increased risk of COVID-19 randomized to low versus moderate dose vitamin D. We hypothesize that moderate dose therapy will reduce rates of COVID-19 compared to low dose therapy because vitamin D will reduce symptomatic infection that prompts testing for COVID-19.

Aim 2: To compare COVID-19 outcomes (symptoms, hospitalization, ICU stay, ventilator use, death) in adults at increased risk of COVID-19 randomized to low vs. moderate dose vitamin D. Consistent with several recent observational analyses, we expect higher doses to improve COVID-19 outcomes.

Subjects will be asked to complete a web-based survey at intake and at 3, 6, 9, and 12 months after enrollment. The intake survey will collect baseline data on subjects' current medications and supplements, sun exposure, exercise, diet and sleep habits, possible COVID-19 symptoms, other influenza-like symptoms, previous exposures to COVID-19, occupation, demographic information, and risks of exposure. The surveys at 3, 6, 9, and 12 months after enrollment will ask the participant or a proxy whether the participant has had a clinically confirmed diagnosis of COVID-19 and the date if so, ask about rates of study medication adherence, and assess for changes in the intake questions about use of other supplements, sun exposure, diet, exercise, and COVID-19 exposures. If the subject reports to have had COVID-19, we will ask about severity, including symptoms, hospitalization and duration, ICU use and duration, need for mechanical ventilation and duration, and death.

ELIGIBILITY:
Inclusion Criteria:

Subjects are able to participate if they:

1. Are 18 years or older.
2. Live in the United States.
3. Are interested in vitamin D as a potential preventive measure against COVID-19 in which they self-administer a daily dose of vitamin D during the 12-month study period.
4. Are willing to complete self-report measures at 5 time points over the course of 12 months by completing a 15-minute survey at intake via web and 10-minute web-based follow-up surveys.

Exclusion Criteria:

Subjects are excluded from study participation if they:

1. Report being pregnant, planning to become pregnant, and/or report breastfeeding during the study period.
2. Report a history of chronic kidney disease, including a history of abnormal GFR and/or creatinine.
3. Report a history of hyperparathyroidism.
4. Report a history of increased falls.
5. Report a history of hypercalcemia.
6. Report a history of gastrointestinal absorptive disorders, including having undergone bariatric surgery.
7. Report a history of kidney stones (1 in past year or 2 in lifetime).
8. Report already taking more than 400 IU of vitamin D daily as recommended by their health care provider, excluding multivitamins and excluding supplements that include vitamin D and calcium together.
9. Report taking D2.
10. Report a history of sarcoidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2093 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Time from randomization to first participant-reported COVID-19 infection | From date of randomization to the earliest of either the first participant-reported COVID-19 infection up to and including 365 days after randomization or right censoring up to 365 days after randomization
  Reported in a post-randomization survey

OTHER OUTCOMES:
COVID-19 infection severity as measured by symptoms using a modified Beat COVID-19 instrument (NCT04337762) | In the first post-randomization survey in which a participant reported COVID-19 infection up to and including 365 days after randomization
  Reported in a post-randomization survey
COVID-19 infection severity as measured by hospital admission | Hospital admissions up to and including 365 days after randomization
  Total number of hospital admissions for COVID-19 infection reported in a post-randomization survey
COVID-19 infection severity as measured by hospitalization with ICU admission | Hospital admissions up to and including 365 days after randomization
  Total number of hospital admissions for COVID-19 infection with an ICU admission reported in a post-randomization survey
COVID-19 infection severity as measured by hospital length of stay | Hospital admissions up to and including 365 days after randomization
  Length of stay for hospital admissions for COVID-19 infection reported in a post-randomization survey
COVID-19 infection severity as measured by ventilator, high-flow nasal oxygen, or helmet-based ventilation | Hospital admissions up to and including 365 days after randomization
  Total number of hospital admissions for COVID-19 infection with ventilator, high-flow nasal oxygen, or helmet-based ventilation reported in a post-randomization survey
COVID-19 infection severity as measured by death | Death up to and including 365 days after randomization
  Notification of study staff

CONTACTS AND LOCATIONS:
Overall Officials: David O Meltzer, MD, PhD, Study Director — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data underlying the text, tables, figures, and appendices of article publications will be made available after deidentification. We will also provide the study protocol and statistical analysis plan. Data will be available six months after article publication until five years following article publication. Researchers wishing to use the data must prepare a protocol for the use of the data which will be reviewed for methodological soundness and potential human subjects concerns by the study investigators and the UChicago Medicine Institutional Review Board. Individual participant meta-analysis and other purposes will be considered. Proposals should be directed to dmeltzer@bsd.uchicago.edu. To gain access, data requestors will need to complete a data access agreement. Data will be accessible through a secure website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available six months after article publication until five years following article publication. The study protocol, SAP, and ICF will be provided to any requesting party. The CSR and analytic code will be provided to any requesting party following publication.
Access Criteria: Researchers wishing to use the data must prepare a protocol for the use of the data which will be reviewed for methodological soundness and potential human subjects concerns by the study investigators and the UChicago Medicine Institutional Review Board. The study protocol, SAP, ICF, CSR and analytic code will be provided to any requesting party.

DOCUMENTS (2):
  • Study Protocol (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT07128069/Prot_001.pdf
  • Statistical Analysis Plan (2025-11-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT07128069/SAP_002.pdf